CLINICAL TRIAL: NCT01508585
Title: Telephone-based Cognitive Behavioral Therapy for Bariatric Surgery Patients: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-0622-BE
Record Dates: First submitted 2011-12-22; First posted 2012-01-12 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Obesity; Eating Disorder
Keywords: Bariatric surgery; Cognitive Behavioral Therapy; Telephone based CBT; Obesity
MeSH Terms: conditions — Obesity; Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pre-Op CBT (Active Comparator): This group will receive CBT (Telephone Based Cognitive Behavioral Therapy) before bariatric surgery
  Interventions: Behavioral: Telephone Based Cognitive Behavioral Therapy
- Post-Op CBT (Active Comparator): This group will receive CBT (Telephone Based Cognitive Behavioral Therapy) after bariatric surgery
  Interventions: Behavioral: Telephone Based Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Telephone Based Cognitive Behavioral Therapy — 6 sessions of Cognitive Behavioral Therapy (CBT), lasting approximately 60 minutes each.
  Other Names: Tele-CBT

SUMMARY:
Bariatric surgery is the most effective treatment for patients with extreme obesity. Psychological interventions are not routinely offered in Bariatric Surgery Programs. Preliminary evidence suggests that Cognitive Behavioral Therapy (CBT) might be effective in reducing binge eating and improving surgical outcomes. The current study will examine whether the addition of telephone-based CBT (Tele-CBT) to the usual standard of care is more effective than the usual standard of care alone, and whether it is more effective when delivered prior to or following bariatric surgery.

DETAILED DESCRIPTION:
Preliminary research suggests that CBT might be effective in reducing eating pathology and improving surgical outcomes.

However, previous studies have examined group-based CBT delivered in person, and most patients cannot feasibly attend weekly therapy appointments at the hospital. Telephone-based CBT offers greater convenience because the service can be delivered during the evening and weekends, and eliminates the need to leave work and travel to hospital appointments. No published studies have examined the effectiveness or feasibility of telephone-based CBT for bariatric surgery patients. This study will examine the effectiveness of Tele-CBT as an adjunctive treatment to the usual standard of care in bariatric surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English
* Have access to telephone and computer with internet access
* Have the capacity to provide informed consent

Exclusion Criteria:

* Active suicidal ideation
* Serious mental illness
* Active severe depression
* Active severe anxiety
* Active post traumatic stress disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2012-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Changes in Depression severity | Baseline, weekly up to 6 weeks and post-intervention, 6 months and 1 year after bariatric surgery
  Measured with "Patient Health Questionnaire" (PHQ-9),a 9-item self-report measure of depression severity
Changes in Anxiety severity | Baseline, post-intervention, 6 months, and one year after bariatric surgery
  Measured by "Generalized Anxiety Disorder Questionnaire" (GAD-7) ,a 7-item self report measure of anxiety severity
Changes in Health-related quality of life | Baseline, post-intervention, 6 months, and one year after bariatric surgery
  Measured by "Short-Form Health Survey" (SF-36), a 36-item self-report measure of health-related quality of life.
Changes in eating pathology | Baseline, post-intervention, 6 months, and 1 year after bariatric surgery
  Measured by the "Binge Eating Scale" (BES) and "Emotional Eating Scale" (EES). The BES is a 16-item self-report measure designed specifically for use with obese individuals that assesses binge eating behaviors as well as associated cognitions and emotions. The EES is a 25-item self-report measure that assesses the tendency to cope with negative affect by eating.

SECONDARY OUTCOMES:
Comparing improvements on the outcome of Tele-CBT before and after bariatric surgery | One year follow-up
  Half the subjects will receive the CBT intervention prior to surgery, and half will receive it after surgery; they will be followed until 1 year post surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Sagar V Parikh, MD, FRCPC, Principal Investigator — University Health Network, Toronto; Raed Hawa, MD,, Study Director — University Health Network, Toronto; Stephanie Cassin, MD, Study Director — University Health Network, Toronto; Susan Wnuk, MD, Study Director — University Health Network, Toronto; Rachel Strimas, Study Director — University Health Network, Toronto; Sanjeev Sockalingam, MD,FRCPC, Study Director — University Health Network, Toronto

REFERENCES:
- [Background] Cassin SE; Sockalingam S; Wnuk S; Strimas R; Royal S; Hawa, R; & Parikh S. Cognitive behavioural therapy for bariatric surgery patients: Preliminary evidence for feasibility, acceptability, and effectiveness. Cognitive and Behavioral Practice 20: 529-543, 2013.